CLINICAL TRIAL: NCT01584401
Title: Temperature Measurement Using a Non Invasive Device
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medisim Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 0295-11-RMC
Record Dates: First submitted 2012-04-22; First posted 2012-04-25 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Body Temperature Measurement
Keywords: Body temperature; Thermometers; Non invasive; Medisim's non invasive thermometers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Main study objectives:

1. To compare the temperature measured using Medisim's thermometers to the temperature measured using mercury or equivalent reference thermometers.
2. To develop more accurate algorithms for measuring on the forehead as well as behind the ear.
3. To test the difference between various forehead measurement locations in order to allow more convenient measuring that is not depended on the exact location.

ELIGIBILITY:
Inclusion Criteria:

* Patients arriving to the emergency room
* A signed consent by the patient or the guardian.

Exclusion Criteria:

* The medical staff decides that patient is not allowed to participate.
* The patient refuses to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Non-blinded, randomized study format. Study population includes 500 patients at all ages and from both genders.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-05

CONTACTS AND LOCATIONS:
Overall Officials: Yehezkel Weissman, Proffessor, Principal Investigator — Schneider Children's Medical Center, Israel
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel